CLINICAL TRIAL: NCT02379741
Title: A First-in-human, Multicenter, Open-label, Multiple Ascending Dose Phase I Study in Patients With Advanced Solid Tumors to Determine the Safety, Pharmacokinetics and Pharmacodynamics of Intratumorally or Intravenously Administered ADC-1013
Brief Title: ADC-1013 First-in-Human Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alligator Bioscience AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-14-1013-C-01
Record Dates: First submitted 2015-02-16; First posted 2015-03-05 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Neoplasms; Solid Tumors
Keywords: Antibodies; Antibodies, Monoclonal; Antineoplastic agent; Physiological effects of drugs; Therapeutic uses; Clinical Trial, Phase I; Immunotherapy, Active; CD40 Antigen; Immunologic Factors; Injections, Intralesional
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — mitazalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADC-1013 intratumoral (Experimental): ADC-1013 (agonistic human monoclonal IgG1 anti-CD40 antibody) administered by intratumoral injection every second week for 8 weeks. Patients that do not progress will be offered continued treatment until complete response, confirmed progressive disease, or clinical deterioration.
  Interventions: Biological: ADC-1013
- ADC-1013 intravenous (Experimental): ADC-1013 (agonistic human monoclonal IgG1 anti-CD40 antibody) administered by intravenous infusion every second week until complete response, confirmed progressive disease, or clinical deterioration.
  Interventions: Biological: ADC-1013

INTERVENTIONS:
Biological: ADC-1013 — Agonistic human monoclonal IgG1 anti-CD40 antibody

SUMMARY:
The purpose of this study is to determine whether ADC-1013 (an agonistic human monoclonal IgG1 anti-CD40 antibody) is safe and tolerable when administered intratumorally (as repeated injections directly into the tumor tissue) or intravenously (as repeated doses directly into a vein) in patients with advanced solid tumors.

ELIGIBILITY:
Major Inclusion Criteria:

* Diagnosis of advanced solid tumor disease
* Performance status of 0-1 on the ECOG scale
* Life expectancy of at least 3 months

Major Exclusion Criteria:

* Organ transplant recipient
* Autoimmune disorder
* Other malignancy (except localized prostate cancer, adequately treated basal skin cancer or carcinoma in-situ of the cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of increasing doses of ADC-1013, assessed by medical review of AE reports and vital signs measurements (blood pressure, pulse rate, body temperature), physical examinations, ECGs and clinical laboratory tests. | From start of study until end of study (appr 28 days after last dose)
  Dose-limiting toxicities (DLTs), maximum tolerated dose (MTD) and recommended Phase 2 dose of ADC-1013 administered intratumorally or intravenously will be defined.

SECONDARY OUTCOMES:
Pharmacokinetics of ADC-1013 after single and repeated administrations assessed by the following parameters: Cmax, Tmax, elimination half-life, AUC0-∞, total serum clearance (CL) and the volume of distribution at steady state (Vss). | From first dose until 55 days after first dose
Immunogenicity of ADC-1013 after repeated administrations assessed by anti-drug antibody (ADA) titers in serum | From first dose until end of study (appr 28 days after last dose)
Clinical efficacy (i.e. anti-tumor activity) of ADC-1013 assessed by immune-related RECIST (irRECIST) and RECIST 1.1. | From start of study until end of study (appr 28 days after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Per Norlén, MD, PhD, Study Director — Alligator Biosciene AB, Sweden; Dorte Nielsen, MD, PhD, Study Chair — Department of Oncology Herlev Hospital, Denmark
Locations (5):
- Center for Cancer Research, Department of Oncology, Herlev Hospital, Herlev, Herlev, Denmark
- Sweden (2):
  - Kliniska prövningsenheten (KPE), Karolinska University Hospital, Solna, Stockholm County
  - Department of Oncology, Uppsala University Hospital, Uppsala, Uppsala County
- United Kingdom (2):
  - Department of Oncology, Queen Elisabeth Hospital, Edgbaston, Birmingham
  - The Clatterbridge Cancer Centre, Bebington, Wirral